CLINICAL TRIAL: NCT00315042
Title: Multinational, Randomized, Double-Blind, Double Dummy, Comparative Study to Evaluate the Efficacy and Safety of 5 Days Telithromycin 25mg/kg od Versus 10 Days Penicillin V 13.3 mg/kg Tid in Children 6 Months to Less Than 13 Years With Streptococcus Pyogenes Tonsillitis/Pharyngitis
Brief Title: TELI TON - Telithromycin in Tonsillitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pediatric development program terminated by sponsor
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6133; HMR3647B/3004
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Tonsillitis; Pharyngitis
Keywords: Tonsillitis; pharyngitis; penicillin; telithromycin; ketolides; clinical trials
MeSH Terms: conditions — Tonsillitis; Pharyngitis | interventions — telithromycin; Penicillins

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Telithromycin (HMR3647)
Drug: Penicillin

SUMMARY:
This is a multinational, randomized (1:1), double blind, double dummy, comparator-controlled, 2 parallel treatment group study in subjects from 6 months to < 13 years of age, with Streptococcus pyogenes tonsillitis/pharyngitis (T/P).Each subject will receive either telithromycin 25 mg/kg once daily for 5 days or penicillin V, 13.3 mg/kg three times daily for 10 days. Matching placebo for telithromycin and penicillin V will also be dispensed for 5 and 10 days respectively, to provide blinding to the different treatment regimens. A positive rapid identification test for streptococcal Group A antigen will be required for all subjects at Visit 1 (Day 1) for entry into the study. Throat swab specimens for bacterial culture, identification, and antibiotic-susceptibility testing will be taken at Visits 1, 3 and 4.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to less than 13 years of age (<13);
* Clinical diagnosis of acute tonsillitis/pharyngitis caused by Streptococcus pyogenes based on:

  * A positive result from a rapid detection throat swab test for Group A streptococcal antigen and submission of a throat swab specimen for bacterial culture, identification, and antibiotic-susceptibility testing; and
  * A sore and scratchy throat and/or pain on swallowing (odynophagia) together with at least 2 of the following clinical signs:

    * Tonsil and/or pharyngeal erythema and/or exudate;
    * Cervical adenopathy;
    * Uvular edema;
    * Fever

Exclusion Criteria:

* Symptoms that collectively suggest nonstreptococcal T/P (eg, laryngitis, coryza, conjunctivitis, diarrhea, cough);
* History of positive throat culture for Streptococcus pyogenes in the absence of clinical signs and symptoms of T/P;
* Infection of the deep tissues of the upper respiratory tract (eg, epiglottitis, retropharyngeal or buccal cellulitis, or abscess of the retropharynx, tonsil, or peritonsillar area) or of the suprapharyngeal respiratory tract and its connecting structures (eg, sinusitis, otitis media, or orbital/periorbital cellulitis);
* History of rheumatic heart disease;
* Females of childbearing potential (ie, have reached menarche);
* Known congenital prolonged QT syndrome;
* Known or suspected uncorrected hypokalemia (≤3 mmol/L [mEq/L]), or hypomagnesemia or bradycardia (<50 bpm);
* Myasthenia gravis;
* Known impaired renal function, as shown by creatinine clearance ≤25 mL/min
* The subject:

  * Is being treated with drugs not permitted by the study protocol ie, cisapride, pimozide, astemizole, terfenadine, ergotamine, dihydroergotamine, Class IA (eg, quinidine and procainamide) or Class III (eg, dofetilide) antiarrhythmic agents, simvastatin, lovastatin and atorvastatin;
  * Is currently being treated with systemic antibacterials or has been treated with systemic antibacterials within 14 days prior to enrollment;- Has been treated with any investigational medication within the last 30 days;
  * Has been treated with rifampicin, phenytoin, carbamazepine, or St. John's wort within the last 2 weeks.
* History of hypersensitivity or intolerance to macrolides, penicillins, or cephalosporins;
* Previous enrollment in this study or previous treatment with telithromycin;
* Children of the investigator or subinvestigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the protocol.

Ages: 6 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 314 (Actual)
Dates: Start 2006-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To compare the bacteriologic efficacy of 5-days of telithromycin to 10-days of penicillin V in subjects at the posttherapy/test-of-cure (TOC) visit in the per protocol population

SECONDARY OUTCOMES:
To compare the bacteriologic efficacy of 5-days of telithromycin to 10-days of penicillin V in subjects at the posttherapy/test-of-cure (TOC) visit andlate posttherapy visit (Visit 4) in the bacteriologic modified intent to treat population

CONTACTS AND LOCATIONS:
Locations (5):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, San Isidro, Buenos Aires, Argentina
- Sanofi-Aventis, Providencia, Santiago Metropolitan, Chile
- Sanofi-Aventis, San José, Costa Rica
- Sanofi-Aventis, Panama City, Panama